CLINICAL TRIAL: NCT03953638
Title: Application of Next Generation Sequencing Technique in Pediatric Bacterial Meningitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Xingtai People's Hospital (Other); Baoding Children's Hospital (Other); Jinan children's hospital (Unknown); Liaocheng People's Hospital (Other); Nanjing Children's Hospital (Other); Shenzhen Baoan Maternal and Child Care Service Centre (Unknown); Jiangxi Children's Hospital (Unknown); Kunming Children's Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Children's Hospital Affiliated to Suzhou University (Unknown)
Responsible Party: Principal Investigator, Gang Liu, Professor, Beijing Children's Hospital
Other Study IDs: 20190514
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Next Generation Sequencing; Pediatric Bacterial Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Cerebrospinal Fluid.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Next Generation Sequencing — To provide rapid etiological diagnosis of patients by means of next-generation sequencing.

SUMMARY:
Pathogen identification is of paramount importance for bacterial meningitis. At present, the pathogen of bacterial meningitis is still mainly based on Gram stain and bacterial culture. However, cerebrospinal fluid (CSF) culture can be negative in children who receive antibiotic treatment prior to CSF examination.Because of the limitations of clinical laboratory testing, more than half of the central nervous system infection cases cannot be clearly diagnosed. The emergence of powerful next-generation sequencing (NGS) technology have enabled unbiased sequencing of biological samples due to its rapid turnaround time. Previous reports highlight the feasibility of applying NGS of CSF as a diagnostic method for central nervous system (CNS) infection. However, the majority of reports are comprised of single case reports and few studies have been reported in the application of NGS for pathogen detection from CSF samples of bacterial meningitis patients, especially in pediatric populations. In this study, we would like to use the NGS technology to detect directly from the CSF samples of children with bacterial meningitis and evaluate the feasibility and significance of the NGS technique on the pathogenic identification of bacterial meningitis.

DETAILED DESCRIPTION:
Bacterial meningitis, also known as purulent meningitis, is caused by a variety of bacterial infections. Although the incidence in infants and children has decreased since the use of conjugated vaccines targeting Haemophilus influenzae type b (Hib), Streptococcus pneumoniae (S. pneumoniae) and Neisseria meningitides (N. meningitides), bacterial meningitis continues to be an important cause of mortality and morbidity in neonates and children throughout the world. The causative pathogens of bacterial meningitis depend on different age of the patient and predisposing factors.

Pathogen identification is of paramount importance for bacterial meningitis. At present, the pathogen of bacterial meningitis is still mainly based on Gram stain and bacterial culture. However, CSF culture can be negative in children who receive antibiotic treatment prior to CSF examination.Because of the limitations of clinical laboratory testing, more than half of the central nervous system infection cases cannot be clearly diagnosed. Although non-culture methods including multiplex PCR and latex agglutination, etc. have been used in clinical microbiology, only one or several specific pathogens could be targeted by these kinds of technology, let alone rare pathogens.

In recent years, the emergence of powerful NGS technology have enabled unbiased sequencing of biological samples due to its rapid turnaround time. Wilson et al presented a case of neuroleptospirosis, resulting in a dramatic clinical improvement with intravenous penicillin after identifying leptospira infection in the CSF by unbiased NGS technology. Unbiased NGS could facilitate identification of all the potential pathogens in a single assay theoretically. Herpes simplex virus1, herpes simplex virus 2 and human herpes virus type 3 were detected using NGS technology from four cases with clinically suspected viral meningoencephalitis respectively. And the results were further validated using polymerase chain reaction (PCR). Further, Yao et al detected Listeria monocytogenes in CSF from three patients with meningoencephalitis by NGS. These reports highlight the feasibility of applying NGS of CSF as a diagnostic method for central nervous system (CNS) infection. However, the majority of reports are comprised of single case reports and few studies have been reported in the application of NGS for pathogen detection from CSF samples of bacterial meningitis patients, especially in pediatric populations. In this study, we would like to use the NGS technology to detect directly from the CSF samples of children with bacterial meningitis and evaluate the feasibility and significance of the NGS technique on the pathogenic identification of bacterial meningitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients highly suspected of bacterial meningitis

Exclusion Criteria:

* Non-bacterial infectious central nervous system (CNS) confirmed by viral meningitis, tuberculous meningitis cryptococcal meningitis and so on
* Autoimmune encephalitis cases
* Central nervous system affected by neoplastic disease
* Hemorrhagic cerebrospinal fluid
* Less than 1ml cerebrospinal fluid
* Refusal to enter the group

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients that are highly suspected of bacterial meningitis.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value (sensitivity and sensibility, positive/negative predictive value) of next-generation sequencing in the pathogen detection of Pediatric Bacterial Meningitis | 2 years
  We aim to collect samples cerebrospinal fluid from patients with Pediatric Bacterial Meningitis. Next-generation sequencing will be performed on the collected samples. Our analysis of the sequencing results will focus on the analysis and identification of pathogen genes and will compare the diagnostic performance of next-generation sequencing with conventional etiological diagnostic methods. We anticipate that next-generation sequencing in Pediatric Bacterial Meningitis will show a greater diagnostic value than the traditional methods (including culture, special pathogen antigen, PCR detection of nucleic acids, etc.).

SECONDARY OUTCOMES:
Diagnostic value (sensitivity and sensibility, positive/negative predictive value) of traditional methods in the pathogen detection of infectious diseases | 2 years
  We aim to collect CSF samples from patients with pediatric bacterial meningitis. Traditional methods including culture, special pathogen serology, PCR detection of nucleic acids, etc, will be performed on the collected samples. Our analysis aims to study the diagnostic power of the traditional diagnostic methods in infectious diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Liu, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No